CLINICAL TRIAL: NCT05181059
Title: Dual-layer Spectral Computerized Tomography for Breast Cancer Detection in Women With Dense Breasts: a Single Centre, Feasibility Study - The DECREAS Study
Brief Title: DLSCT for Breast Cancer Detection in Women With Dense Breasts
Acronym: DECREAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NL76792.091.21
Record Dates: First submitted 2021-12-16; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Breast Neoplasms; Breast Density; Radiographic Image Interpretation, Computer-Assisted
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dual-layer spectral computerized tomography (DLSCT) — Contrast enhanced DLSCT scan using a 128-slice dual-layer detector (IQon Spectral CT, Philips Health Systems) will be performed. Patients will be placed in prone position during the DLSCT scan in order to improve the visualisation of breast tissue and comparability with MRI images. During the examination we will administer a nonionic low-osmolar iodinated contrast agent (Optiray©) in order to visualise tumor angiogenesis.

SUMMARY:
The main objective of this project is to demonstrate the feasibility of DLSCT to detect breast cancer in women with dense breasts.

Patients with locoregional advanced primary breast cancer and heterogeneously (n = 7) or extremely dense breasts (n = 7) as determined by mammography will be included in this study. These patients have an indication for a positron emission tomography computed tomography (PET-CT) scan to search for distant metastases. In this study the participants will undergo an additional contrast enhanced DLSCT scan to determine the feasibility of spectral CT to detect breast cancer in women with dense breasts.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histopathologically proven locoregional advanced primary breast cancer:

  1. Tumors > 5 cm (= T3) or
  2. Tumors with invasion of the skin or chest wall (= T4) or
  3. Any tumor with ≥ 4 axillary lymph nodes or ipsilateral internal mammary, infraclavicular or supraclavicular nodal involvement (= N2-3)
* Heterogeneously or extremely dense breasts as described by visual assessment on full-field digital mammograms: category C or D according to the ACR BI-RADS lexicon

Exclusion Criteria:

* History of allergic reactions to iodinated contrast agents
* Pregnancy or breast feeding
* Treatment of thyroid disease with radioactive iodine
* Use of metformin
* Creatinine clearance < 45 ml/min
* Chronic or acutely worsening renal disease
* Patients who are declared incompetent

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Secondary care clinic
Sampling Method: Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Visual tumor conspicuity | On the same 1 day as the regular PET-CT scan was performed
  The conspicuity of tumors will be graded on a 4-point confidence scale
BI-RADS score | On the same 1 day as the regular PET-CT scan was performed
  BI-RADS score according to the ACR BI-RADS lexicon

SECONDARY OUTCOMES:
Iodine enhancement | On the same 1 day as the regular PET-CT scan was performed
  Iodine enhancement will be measured in Hounsfield Units (HU).
Iodine content | On the same 1 day as the regular PET-CT scan was performed
  Iodine content will be measured mg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Laura N Deden, Principal Investigator — Rijnstate Hospital; Maxime V.P. Schyns, MD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands